CLINICAL TRIAL: NCT03580837
Title: Breast MRI for Neaodjuvant Chemotherapy Response Prediction and Evaluation in Breast Cancer, With Focus on Background Parenchymal Enhancement
Brief Title: Breast MRI for Neaodjuvant Chemotherapy Response Prediction and Evaluation in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6788
Record Dates: First submitted 2018-01-03; First posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this retrospective study is to evaluate the value of pre-treatment and post-treatment multimodality MRI study, including quantitative evaluation of background parenchymal enhancement, for response prediction and evaluation. This study will include 100 patients treated in a single institution between 2011 and 2016

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients with breast cancer treated with neoadjuvant chemotherapy
* Patients with pre- and post-chemotherapy MRI
* Patients who have given their agreement to use their data for research purposes.

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer treated with neoadjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of of pathologic enhancement of breast by MRI | 1 hour after the realization of the MRI
  This work concerns 110 patients treated with neoadjuvant chemotherapy for breast cancer and having received a breast MRI in pre and post-chemiotherapy at the Hautepierre Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien MOLIERE, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service Imagerie 1, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No